CLINICAL TRIAL: NCT07002177
Title: An Open-label, Multicenter, Phase Ib/II Clinical Study to Evaluate the Safety and Efficacy of Multiple Combination Therapies With FWD1802 in Subjects With ER-positive/HER2-negative Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: A Phase Ib/II Study to Evaluate Multiple Combination Therapies of FWD1802 in Patients With ER+/HER2- BC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forward Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWD1802-002C
Record Dates: First submitted 2025-05-14; First posted 2025-06-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Locally Advanced Breast Cancer (LABC); ER+ Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; ribociclib; Tablets; abemaciclib; Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FWD1802 in combination with Palbociclib (CDK4/6 inhibitor) with or without LHRH agonist； (Experimental)
  Interventions: Drug: FWD1802; Drug: Palbociclib 125mg
- FWD1802 in combination with Ribociclib (CDK4/6 inhibitor) with or without LHRH agonist (Experimental)
  Interventions: Drug: FWD1802; Drug: Ribociclib 200Mg Oral Tablet
- FWD1802 in combination with Abemaciclib (CDK4/6 inhibitor) with or without LHRH agonist (Experimental)
  Interventions: Drug: FWD1802; Drug: Abemaciclib 150 MG
- FWD1802 in combination with Everolimus (mTOR inhibitor) with or without LHRH agonist (Experimental)
  Interventions: Drug: FWD1802; Drug: Everolimus 10 mg

INTERVENTIONS:
Drug: FWD1802 — orally QD with 28 days each cycle, treatment till disease progression or intolerable toxicity or withdraw for other reasons
Drug: Palbociclib 125mg — Dose: 125 mg Route: Orally Frequency: Once daily (QD) Schedule: Administered for 21 consecutive days, followed by a 7-day treatment break (3-weeks-on/1-week-off), constituting a 28-day cycle
  Arms: FWD1802 in combination with Palbociclib (CDK4/6 inhibitor) with or without LHRH agonist；
Drug: Ribociclib 200Mg Oral Tablet — Dose: 600 mg Route: Orally Frequency: Once daily (QD) Schedule: Administered for 21 consecutive days, followed by a 7-day treatment break, constituting a 28-day cycle
  Arms: FWD1802 in combination with Ribociclib (CDK4/6 inhibitor) with or without LHRH agonist
Drug: Abemaciclib 150 MG — Dose: 150 mg Route: Orally Frequency: BID Schedule: Everyday
  Arms: FWD1802 in combination with Abemaciclib (CDK4/6 inhibitor) with or without LHRH agonist
Drug: Everolimus 10 mg — Dose: 10 mg Route: Orally Frequency: QD Schedule: Everyday
  Arms: FWD1802 in combination with Everolimus (mTOR inhibitor) with or without LHRH agonist

SUMMARY:
This is a Study to Evaluate the Efficacy and Safety of Multiple Combination Therapies with FWD1802 in Subjects with ER-positive/HER2-negative Unresectable Locally Advanced or Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Subjects consent to provide blood samples for centralized laboratory testing of ESR1 mutation status and other biomarkers.
* Histologically or cytologically confirmed ER-positive/HER2-negative locally advanced or metastatic breast cancer
* Subjects must meet at least one of the following criteria: postmenopausal or prior bilateral oophorectomy, or postmenopausal or Premenopausal/perimenopausal women must agree to receive and maintain approved luteinizing hormone-releasing hormone (LHRH) agonist therapy during study treatment
* Prior Therapy Requirements:Subjects must meet all of the following criteria:

  1. Progression during/after, intolerance to, ineligibility for, or refusal of standard therapy
  2. Endocrine therapy history:

     Recurrence during or within 1 year after completing ≥2 years of adjuvant endocrine therapy;OR progression after ≥1 line of endocrine therapy for advanced breast cancer(ABC) with ≥6 months of maintenance therapy (no restriction on the number of prior endocrine therapy lines).
  3. ≤2 prior lines of chemotherapy for ABC
  4. No prior SERD (selective estrogen receptor degrader) therapy except fulvestrant
  5. Everolimus combination arm: Prior CDK4/6 inhibitor therapy requiredf) CDK4/6 inhibitor combination arm:Permitted ≤1 line of prior non-investigational CDK4/6 inhibitor therapy;If only received adjuvant CDK4/6 inhibitor therapy, recurrence must occur >12 months after treatment completion Note: Antibody-drug conjugates (ADCs) are classified as chemotherapy in this study.
* Phase Ib: At least one evaluable lesion per RECIST v1.1, allowed subjects with osteolytic bone lesion(s) confirmed by CT/MRI.Phase II: At least one measurable lesion per RECIST v1.1.

Subject must have sufficient organ and bone marrow functions at screening.

Exclusion Criteria:

* Leptomeningeal metastasis (carcinomatous meningitis)；Spinal cord compression；Symptomatic or clinically unstable central nervous system (CNS) metastases；
* History or any persistent chronic gastrointestinal disorders or other conditions of impaired absorption that may interfere with oral absorption of the investigational drug
* Symptomatic visceral metastases , or clinically symptomatic and unstable effusions;Pleural effusion;Ascites;Pericardial effusion or Pulmonary lymphangitis carcinomatosa. Prior intracavitary infusion therapy should have more than 14 days of stabilization,
* Prior therapy with any selective estrogen receptor degrader (SERD) or similar agents other than fulvestrant
* Inadequate washout period for prior anticancer therapies.
* Type 1 diabetes mellitus; Type 2 diabetes mellitus with poor glycemic control at screening(applies only to the everolimus combination arm).
* Subjects will be excluded if they meet any of the following:

  1. Interstitial lung disease or drug-induced ILD history, OR evidence of active pneumonitis on chest CT scan within 4 weeks prior to first study treatment.
  2. Severe pulmonary disease at screening, including but not limited to:Severe asthma;Severe chronic obstructive pulmonary disease (COPD) Idiopathic
* Uncontrolled hypertension despite antihypertensive therapy, defined as:Systolic blood pressure (SBP) >150 mmHg OR Diastolic blood pressure (DBP) >95 mmHg.
* Active cardiac disease or history of cardiac dysfunction

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 196 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ib- Dose-Limiting Toxicity (DLT). | Approximately 1.5 years
Phase Ib- Maximum Tolerated Dose (MTD). | Approximately 1.5 years
Phase Ib- Recommended Phase II Dose (RP2D). | Approximately 1.5 years
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Approximately 2 years
  Number and proportion of participants experiencing any treatment-emergent adverse event during the study period.
  Assessment criteria: Events will be categorized as "related" or "unrelated" to study drug based on investigator's causality assessment.
  Reporting format: Frequency counts and percentages stratified by severity grade (Grade 1-5 as per NCI-CTCAE v5.0).
Severity Grading of Adverse Events | Approximately 2 years
  Maximum severity grade of treatment-emergent adverse events experienced by participants.
  Assessment tool: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
  Reporting format: Proportion of participants with events in each severity category (Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening; Grade 5=death).
Clinically Significant Abnormalities in 12-Lead ECG Parameters | Approximately 2 years
  Number of participants with clinically significant changes in electrocardiogram parameters from baseline.
  Assessed parameters: QTc interval, PR interval, QRS duration, heart rate.
Vital Sign Abnormalities | Approximately 2 years
  Proportion of participants with clinically significant deviations in vital signs:
  Parameters: Systolic/diastolic blood pressure (mmHg), heart rate (bpm), respiratory rate (breaths/min), body temperature (°C).
Serious Adverse Events (SAEs) Incidence | Approximately 2 years
Phase II- Investigator-assessed Objective Response Rate (ORR) based on RECIST v1.1. | Approximately 2 years

SECONDARY OUTCOMES:
Phase Ib- PK Assessment-Tmax | Approximately 1.5 years
  Time to Cmax (Tmax).
Phase Ib- PK Assessment-Cmax | Approximately 1.5 years
  Maximum plasma concentration (Cmax)
Phase Ib- PK Assessment-AUC0-t | Approximately 1.5 years
  Area under the concentration versus time curve from time 0 to the last measurable concentration (AUC0-t)
Phase Ib- PK Assessment-AUC0-inf | Approximately 1.5 years
  The area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf)
Phase Ib- PK Assessment-t1/2 | Approximately 1.5 years
  elimination half-life time (t1/2)
Efficacy Assessment-ORR | Approximately 2 years
  Tumor response assessments by the corresponding criteria by RECIST v1.1 to assess Objective response rate (ORR)
Efficacy Assessment-CBR | Approximately 2 years
  Clinical benefit rate (CBR)
Efficacy Assessment-DOR | Approximately 2 years
  Duration of response (DoR）
Efficacy Assessment-DCR | Approximately 1.5 years
  Disease control rate (DCR)
Efficacy Assessment-PFS | Approximately 2 years
  Progression-free survival (PFS) by IRC according to RECIST 1.1.PFS is defined as time from the first dose until disease progression or death from any cause, whichever occurs first.
Efficacy Assessment-OS | Approximately 2 years
  Overall survival (OS).OS is defined as time from date of the first dose to date of death due to any cause.
Pharmacokinetic (PK) Parameters:Plasma Concentration at Each Sampling Time Point. | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai, China